CLINICAL TRIAL: NCT02618421
Title: A Cross-sectional Population Representative Internet Survey to Estimate Prevalence of Lower Urinary Tract Symptoms (LUTS) in China, Taiwan and South Korea
Brief Title: A Cross-sectional Internet Survey to Estimate Prevalence of Lower Urinary Tract Symptoms (LUTS)
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Singapore Pte. Ltd. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: URO-MA-1006
Record Dates: First submitted 2015-11-26; First posted 2015-12-01 (Estimated); Last update posted 2024-10-22 (Actual); Status verified 2019-01

CONDITIONS: Lower Urinary Tract Symptoms
MeSH Terms: conditions — Lower Urinary Tract Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants Aged 40 Years or Over: Cross-section of general population of males and females in China, Taiwan, and South Korea

SUMMARY:
The purpose of the study is to determine prevalence of lower urinary tract symptoms in population aged 40 years or over, in China, Taiwan and South Korea using latest ICS definition.

DETAILED DESCRIPTION:
The research question for this study pertains to assessing prevalence and symptom specific bother of LUTS and its impact on HRQL, work productivity, mental and sexual health across China, Taiwan and South Korea, using latest ICS definition.

The research is a cross sectional population-representative internet survey among general population of males and females aged 40 years or older. The research would be an internet-based self-administration survey across China, Taiwan and South Korea.

The primary objective of the study is to determine the prevalence of lower urinary tract symptoms in population aged 40 years or over, in China, Taiwan and South Korea using latest ICS definition.

Secondary objectives of the study are:

* To examine the symptom-specific bother of LUTS
* To evaluate impact of these symptoms on health-related quality of life, work productivity, mental and sexual health using standard survey instruments
* To explore the differences in prevalence of LUTS across males and females, across age groups, across different socioeconomic strata and across China, Taiwan and South Korea
* To examine the extent of overlap of voiding and storage symptoms among the study participants
* To explore treatment seeking behavior and determine treatment rate and satisfaction with current treatment

ELIGIBILITY:
Inclusion Criteria:

* Aged 40 years or older on the date of survey
* Able to read local language
* Able to access the internet and use a computer (with or without the help of an assisting person who may or may not be a family member)
* Provides of informed consent

Exclusion Criteria:

* Is pregnant
* Diagnosed as having urinary tract infection by a physician in the past one month which may be cured or persisting

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population aged 40 years or over, in China, Taiwan and South Korea
Sampling Method: Probability Sample
Enrollment: 8284 (Actual)
Dates: Start 2015-06-02 (Actual); Primary Completion 2015-07-20 (Actual); Study Completion 2015-07-20 (Actual)

PRIMARY OUTCOMES:
The prevalence of lower urinary tract symptoms using ICS 2002 symptom definition | At enrollment
  Prevalence of lower urinary tract symptoms in population aged 40 years or over, in China, Taiwan and South Korea using ICS 2002 symptom definition. Measured at enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Singapore

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Chow PM, Chuang YC, Hsu KCP, Shen YC, Liu SP. Impact of Female Stress Urinary Incontinence on Quality of Life, Mental Health, Work Limitation, and Healthcare Seeking in China, Taiwan, and South Korea (LUTS Asia): Results from a Cross-Sectional, Population-Based Study. Int J Womens Health. 2022 Dec 28;14:1871-1880. doi: 10.2147/IJWH.S383651. eCollection 2022. PMID 36597480
- [Derived] Cheng MC, Liu SP, Chuang YC, Hsu KCP, Chow PM. Prevalence and impacts of male urinary incontinence on quality of life, mental health, work limitation, and health care seeking in China, Taiwan, and South Korea (LUTS Asia): Results from a cross-sectional, population-based study. Investig Clin Urol. 2022 Jan;63(1):71-82. doi: 10.4111/icu.20210259. PMID 34983125
- [Derived] Wang JY, Liao L, Liu M, Sumarsono B, Cong M. Epidemiology of lower urinary tract symptoms in a cross-sectional, population-based study: The status in China. Medicine (Baltimore). 2018 Aug;97(34):e11554. doi: 10.1097/MD.0000000000011554. PMID 30142751
- [Derived] Chow PM, Liu SP, Chuang YC, Lee KS, Yoo TK, Liao L, Wang JY, Liu M, Sumarsono B, Jong JJ. The prevalence and risk factors of nocturia in China, South Korea, and Taiwan: results from a cross-sectional, population-based study. World J Urol. 2018 Nov;36(11):1853-1862. doi: 10.1007/s00345-018-2329-0. Epub 2018 May 23. PMID 29796775
- [Derived] Liu SP, Chuang YC, Sumarsono B, Chang HC. The prevalence and bother of lower urinary tract symptoms in men and women aged 40 years or over in Taiwan. J Formos Med Assoc. 2019 Jan;118(1 Pt 1):170-178. doi: 10.1016/j.jfma.2018.03.006. Epub 2018 Apr 11. PMID 29655606
- [Derived] Lee KS, Yoo TK, Liao L, Wang J, Chuang YC, Liu SP, Chu R, Sumarsono B. Association of lower urinary tract symptoms and OAB severity with quality of life and mental health in China, Taiwan and South Korea: results from a cross-sectional, population-based study. BMC Urol. 2017 Nov 21;17(1):108. doi: 10.1186/s12894-017-0294-3. PMID 29162085
- [Derived] Chapple C, Castro-Diaz D, Chuang YC, Lee KS, Liao L, Liu SP, Wang J, Yoo TK, Chu R, Sumarsono B. Prevalence of Lower Urinary Tract Symptoms in China, Taiwan, and South Korea: Results from a Cross-Sectional, Population-Based Study. Adv Ther. 2017 Aug;34(8):1953-1965. doi: 10.1007/s12325-017-0577-9. Epub 2017 Jul 7. PMID 28687936